CLINICAL TRIAL: NCT00384241
Title: Inflammatory Factors, Genes and Stress Induced Pressure Natriuresis in Youth
Brief Title: Evaluating the Relationship Between Inflammation, Genetics, and Stress in the Development of High Blood Pressure
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1359; R21HL085817 (NIH); 1R21HL085817-01 (NIH)
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Hypertension
Keywords: Blood Pressure, High; Stress; Inflammation
MeSH Terms: conditions — Hypertension; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples of 500 subjects have been collected and stored in previous funded studies.
  Buccal swabs from 599 biological parents have been collected from the current study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children: Children age 15-19, self reported as African American of European Origin, healthy non-smoker, with normal blood pressure, exposed to an activity to that results in induced stress
  Interventions: Behavioral: Induced Stress
- Parents: Collection of buccal swab Parent of participants in the Children Arm
  Interventions: Procedure: Buccal Swab

INTERVENTIONS:
Behavioral: Induced Stress — Participation in an active coping task by playing a video game against another participant.
  Groups: Children
Procedure: Buccal Swab — One Buccal swab collected from each parent
  Groups: Parents

SUMMARY:
High blood pressure affects nearly one third of all individuals in the United States. If left untreated, it can lead to stroke, heart failure, heart attack, kidney failure, or blindness. For many people, the exact cause of high blood pressure is unknown, but it is believed that both genetic and environmental factors contribute to the development of the condition. The purpose of this study is to examine the importance of genetics, inflammation, and stress on the development of high blood pressure.

DETAILED DESCRIPTION:
High blood pressure is a complex condition that can be caused by many factors, including obesity, diet, genetics, or stress. Maintaining a healthy balance of sodium in the body is important for adequate blood pressure control. Some individuals experience sustained high blood pressure during periods of extended stress, combined with the inability to excrete enough sodium through urine to re-establish normal blood pressure levels. This type of stress-induced high blood pressure is related to interleukin-6 (IL-6), a protein that stimulates inflammation and immune responses. To determine the interaction between stress, inflammation, and genetics, this study will examine the role of IL-6 in regulating sodium levels and blood pressure in individuals undergoing stress. This information will be useful in determining new ways to evaluate risk factors for high blood pressure.

This study will examine previously collected DNA samples from young adults who participated in prior genetic studies. There will be no study visits for participants. IL-6, IL-6R, glycoprotein 130 (gp130), and C-reactive protein (CRP) genes will be analyzed in all samples; changes in plasma levels of IL-6 and CRP in response to stress will be examined in selected samples. The parents of participants will be asked to provide cheek swabs for additional DNA analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participated in two previous NIH funded studies HL073260, HL077230
* Biological parents willing to participate in the study
* African American or European origins

Exclusion Criteria:

* Non-biological parents

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 15-19 years old African American and European American school children.
Sampling Method: Non-Probability Sample
Enrollment: 1099 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Zhu, MD, PhD, Principal Investigator — Augusta University
Locations (1):
- Medical College of Georgia, Georgia Regents University, Augusta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A study record search was completed on 500 youth for inflammatory marker Interleukin 6 (IL-6), genetic polymorphism and stress induced urinary sodium secretion data. 599 parents of identified subjects were asked to submit Buccal swabs for the analysis of IL-6 genes.
Groups:
- Children: Genotyping and IL-6 levels of 500 children enrolled in two previous studies were collected in the current study. Other phenotype data: Baseline blood pressure, stress blood pressure, and recovery blood pressure; Baseline stress and recovery urinary sodium excretion that were collected in two previous studies were utilized in the current study.
- Parents: Buccal swabs from the Parents of 500 subjects in the children arm were collected and analyzed for genetic variations. Some parents submitted duplicate swabs if more than 1 child was represented in the 500 subjects.
Period: Overall Study
Arm/Group | Children | Parents
Started | 500 | 599
Completed | 500 | 599
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Children: African American and Caucasian children age 15-19.
- Parents: African American and Caucasian parents, age 18-65.
- Total: Total of all reporting groups
Arm/Group | Children | Parents | Total
Number analyzed (Participants) | 500 | 599 | 1099
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 500 | 0 | 500
  Between 18 and 65 years | 0 | 599 | 599
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 457 | 693
  Male | 264 | 142 | 406
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 250 | 389 | 639
  White | 250 | 210 | 460
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary Sodium Excretion (UNaV)
Description: The value of Stress induced UNaV as determined by delta UNaV = stress UNaV - baseline UNaV.
Time Frame: Baseline and 4 hour
Population: All 500 subjects in the group Children were analyzed. This data was not intended to be analyzed for Arm 2 Parents.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Children: 500 children age 15-19, self reported as African American or of European origin, healthy, non-smoker with normal blood pressure that participated in two previous studies
Arm/Group | Children
Number analyzed (Participants) | 500
pg/ml
  Baseline | 11.8 (5.6)
  4 hours | 15.2 (7)

2. Secondary Outcome: The Effect of Change in Stress Induced IL-6 on Systolic Blood Pressure
Description: Stress induced systolic blood pressure (SBP) data generated from two previous studies was collected. In the previous studies, systolic blood pressures were measured before and after completing a video game challenge. Stress induced SBP is defined as delta SBP = stress SBP - baseline SBP.
Time Frame: baseline and 4 hours
Population: All 500 subjects in the group Children were analyzed. This data was not intended to be analyzed for Arm 2 Parents.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Children
Number analyzed (Participants) | 500
mmHg
  Baseline | 108.9 (10.1)
  4 hours | 113.3 (11.9)

ADVERSE EVENTS:
Groups:
- Children: African American and Caucasian children age 15 - 19.
- Parents: African American and Caucasian parents age 18 - 65
Arm/Group | Children | Parents
Serious Adverse Events (participants affected / at risk) | 0/500 | 0/599
Other Adverse Events (participants affected / at risk) | 0/500 | 0/599

LIMITATIONS AND CAVEATS:
No treatment was given.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No